CLINICAL TRIAL: NCT04133077
Title: A Prospective Study of Xenografts Development from Samples Taken from Surgical Specimens of Patients with Triple Negative or Luminal B Breast Cancer
Brief Title: Xenografts Development from Surgical Tumor Samples of Patients with Triple Negative or Luminal B Breast Cancer
Acronym: XenoBreast
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Jean Perrin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2020-A00398-31
Record Dates: First submitted 2019-10-16; First posted 2019-10-21 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer Female
Keywords: PDX

STUDY DESIGN:
Intervention Model Description: The intervention consists in the realization of additional blood samples to carry out serologies and genetic analyses
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Succeed PDX (Other): Genetic analysis will be performed in patients who got a successful PDX
  Interventions: Biological: blood samples collection

INTERVENTIONS:
Biological: blood samples collection — Serology and genetic analyses will be performed in patients blood samples

SUMMARY:
Patient derived xenografts (PDX) from mammary tumors are usually made from metastatic tumors. Indeed, PDX from primitive mammary tumors or after neoadjuvant treatment are still rare. However, the realization of such PDX (from primitive mammary tumors or after neoadjuvant treatment) would make it possible to have a better knowledge of the tumor heterogeneity to the therapeutic response, to explore the models of tumor evolution during metastatic progression and also observe the mechanisms of tumor resistance in the case of non-metastatic tumors. It therefore seems necessary to develop PDX from primitive tumors in order to observe firstly the success rate of PDX; on the other hand, the drift of the initial heterogeneity, measured by comparison of the histomolecular profile of the tumors with that of the PDXs. It aims to develop xenografts from tumor samples from surgical specimens of patients with triple negative or luminal B breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* ECOG (Eastern Cooperative Oncology Group) performance status ≤ 2
* Signature of the participation consent to the study,
* Affiliation to a social security scheme
* Major woman with:

  * metastatic triple-negative (TN) breast cancer, histologically proven before treatment and high grade, receiving neoadjuvant chemotherapy and having, after treatment, a breast residue of at least 15 mm on the specimen. The mammary residue will measure at least 15 mm on the mammography performed at the end of neoadjuvant treatment
  * metaplastic triple-negative (TN) breast cancer, histologically proven before treatment and high grade, treated by primary surgery with a tumor size of at least 15 mm on the specimen.
  * an inflammatory TN breast cancer (T4d), histologically proven prior to treatment, receiving neoadjuvant chemotherapy and having, after treatment, a breast residue of at least 15 mm on the specimen. The mammary residue will measure at least 15 mm on the mammography performed at the end of the neoadjuvant treatment.
  * non-metaplastic or inflammatory TN breast cancer, histologically proven prior to treatment, receiving neoadjuvant chemotherapy and having, after treatment, a mammary residue of at least 30 mm on the specimen. The mammary residue will measure at least 15 mm on the mammography performed at the end of the neoadjuvant treatment.
  * Luminal B breast cancer (LB), histologically proven prior to treatment, receiving neoadjuvant chemotherapy and having, after treatment, a mammary residue of at least 30 mm on the specimen. The mammary residue will measure at least 15 mm on the mammography performed at the end of the neoadjuvant treatment.
  * histologically proven metastatic TN or metastatic breast cancer with an operable metastasis whose residual size, after chemotherapy, is at least 10 mm on the specimen. Residual metastasis will be at least 15 mm on imaging.
* Patients in a metastatic situation can be included regardless of the therapeutic line.

Exclusion Criteria:

* Pregnant woman
* Patient deprived of liberty by court or administrative decision
* In neoadjuvant situation: no neoadjuvant treatment by radiotherapy or hormone therapy
* Refusal to participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2021-11-19 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of successfull PDX | 2 years
  PDX will be realized from patient tumor by transplanting a small fragment in a nude mouse. Once the tumor is enough grown up, the tumor is extracted to repeat this step 3 times until we get the fourth PDX with a successful tumor growth.

SECONDARY OUTCOMES:
Histological subtype | 2 years and 4 months
  Comparaison of initial tumor histological subtype with PDX histological subtype
expression of estrogen receptors | 2 years and 4 months
  Comparaison of initial tumor expression of estrogen receptors with PDX expression of estrogen receptors
expression of progesterone receptors | 2 years and 4 months
  Comparaison of initial tumor expression of progesterone receptors with PDX expression of progesterone receptors
status of the amplification of the ERBB2 gene | 2 years and 4 months
  Comparaison of initial tumor's ERBB2 gene amplification status with PDX's ERBB2 gene amplification status
expression of androgen receptors | 2 years and 4 months
  Comparaison of initial tumor expression of androgen receptors with PDX expression of androgen receptors
tumor molecular classification | 2 years and 4 months
  Comparaison of initial tumor molecular expression with PDX molecular classification (luminal A, luminal B, HER2 enriched or triple negative)
Exome sequencing | 2 years and 4 months
  Comparaison of genetic alterations between intial tumor, PDX and blood sample

CONTACTS AND LOCATIONS:
Overall Officials: Xavier DURANDO, Professor, Principal Investigator — Centre Jean Perrin
Locations (1):
- Centre Jean PERRIN, Clermont-Ferrand, Puy-de-Dôme, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Veyssiere H, Passildas J, Ginzac A, Lusho S, Bidet Y, Molnar I, Bernadach M, Cavaille M, Radosevic-Robin N, Durando X. XENOBREAST Trial: A prospective study of xenografts establishment from surgical specimens of patients with triple negative or luminal b breast cancer. F1000Res. 2020 Oct 9;9:1219. doi: 10.12688/f1000research.26873.3. eCollection 2020. PMID 34249349